CLINICAL TRIAL: NCT06006702
Title: A Phase 1, Multi-cohort, Open-label Study to Evaluate the Relative Bioavailability of Capsule and Tablet Formulations of TYRA-300-B01, and to Evaluate the Safety, Tolerability, and Food Effect of TYRA-300-B01 Tablets in Healthy Adult Participants
Brief Title: A Relative Bioavailability and Food Effect Study of TYRA-300-B01 Capsule and Tablet Formulations in Healthy Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TYR300-102
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bioavailability Tablet vs Capsule Formulation (Experimental): TYRA-300-B01 single oral dose of tablet or capsule crossover followed by twice-daily tablet dosing
  Interventions: Drug: TYRA-300-B01
- Food Effect Tablet Formulation (Experimental): TYRA-300-B01 single oral dose of tablet in the fed and fasted state
  Interventions: Drug: TYRA-300-B01
- Pharmacokinetic Tablet Formulation (Experimental): TYRA-300-B01 single oral dose
  Interventions: Drug: TYRA-300-B01
- Pharmacokinetic Mini-Tablet Formulation (Experimental): TYRA-300-B01 multiple-dose mini-tablet formulation
  Interventions: Drug: TYRA-300-B01

INTERVENTIONS:
Drug: TYRA-300-B01 — TYRA-300 is an oral, novel potent FGFR 3-selective tyrosine kinase inhibitor that targets tumors that contain activating gene alterations of FGFR3.

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of capsule and tablet formulations of TYRA-300-B01, and to evaluate the safety, tolerability, and food effect of TYRA-300-B01 tablets in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, multi-cohort trial studying TYRA-300-B01, a novel, potent fibroblast growth factor receptor (FGFR) 3-selective tyrosine kinase inhibitor, in healthy, adult participants. The purpose of this study is to evaluate the relative bioavailability of capsule and tablet formulations of TYRA-300-B01, and to evaluate the safety, tolerability, and food effect of TYRA-300-B01 tablets in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential, between 18 and 55 years of age
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory assessments
* Body mass index (BMI) 18 to 32 kg/m^2 (inclusive)
* Cohorts 1 and 2 ethnicity requirements: none
* Cohort 3 ethnicity requirements: first- or second-generation Japanese participants

Exclusion Criteria:

* Significant history of any hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, immunologic, musculoskeletal disease, or allergic disease (as determined by the Investigator)
* Any ocular condition likely to increase the risk of eye toxicity
* Gastrointestinal disorders that will affect oral administration or absorption of TYRA-300-B01
* Females of child-bearing potential and males who plan to father a child while enrolled in this study

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics single-dose Cmax | Up to 48 hours post-dose
  maximum plasma concentration (Cmax)
Pharmacokinetics multiple-dose Cmax | Up to 24 hours post-dose
  maximum steady-state plasma concentration (Cmax)
Pharmacokinetics multiple-dose Cmin | Up to 24 hours post-dose
  average steady-state trough plasma concentration (Cmin)
Pharmacokinetics single dose Tmax | Up to 48 hours post-dose
  time to reach maximum plasma concentration (Tmax)
Pharmacokinetics single and multiple dose AUC | Up to 48 hours post-dose
  area under the plasma concentration-time curve (AUC)
Pharmacokinetics single dose CL/F | Up to 48 hours post-dose
  apparent total clearance (CL/F)
Pharmacokinetics single dose Vz/F | Up to 48 hours post-dose
  apparent volume of distribution (Vz/F)
Pharmacokinetics single dose t1/2 | Up to 48 hours post-dose
  half-life of TYRA-300
Pharmacokinetics multiple-dose RCmax | Up to 24 hours post-dose
  accumulation ratio for Cmax (RCmax)
Pharmacokinetics multiple-dose RAUC | Up to 24 hours post-dose
  accumulation ratio for AUC

SECONDARY OUTCOMES:
Safety and tolerability | Initiation of study treatment up to 7-days post treatment
  number of participants with adverse events (AEs), serious adverse events (SAEs), adverse events of special interest (AESIs) as a measure of safety and tolerability
Safety and tolerability | Initiation of study treatment up to 7-days post treatment
  Frequency in changes in laboratory parameters and physical signs of toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Doug Warner, M.D., Study Chair — Tyra Biosciences, Inc
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia